CLINICAL TRIAL: NCT04964674
Title: Psychometric Testing and Cue Utilization During Cued Visual Search
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Attempts at online data collection led to poor data quality (many missing data points from one task of the set). Study was terminated, given the data quality issues.
Sponsor: Lehigh University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1R15EY030247-01A1 (NIH)
Record Dates: First submitted 2021-04-14; First posted 2021-07-16 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Healthy
Keywords: attention; visual search

STUDY DESIGN:
Intervention Model Description: Within-subjects measures, individual differences analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Attentional Tests- Miyake and others (Experimental): All participants will complete a series of behavioral tasks, including cued visual search with positive, negative, and neutral cues, Miyake executive attention tasks, and a visual working memory task. Single Arm.
  Interventions: Behavioral: Behavioral Measurement

INTERVENTIONS:
Behavioral: Behavioral Measurement — Take measurements of behavioral performance

SUMMARY:
The experimenters will examine the relationship between utilization of positive (target cue) and negative (distractor cue) templates during a cued visual search task with performance on a set of measures related to executive functions associated with attentional control: shifting, updating, and inhibition.

DETAILED DESCRIPTION:
The experimenters will utilize the typical procedures for the cued attentional task, while also deploying the Miyake executive function analysis. Data will also include a working memory capacity measure.

ELIGIBILITY:
Inclusion Criteria:

* Normal or corrected-to-normal visual acuity, normal color vision

Exclusion Criteria:

* age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-08-27 (Actual); Study Completion 2022-08-27 (Actual)

PRIMARY OUTCOMES:
Positive, Negative, Neutral Attention Task Performance Speed | 1 day
  Reaction times on visual search task with positive, negative, and neutral cues
Positive, Negative, Neutral Attention Task Performance Accuracy | 1 day
  Accuracy on visual search task with positive, negative, and neutral cues
Miyake Executive Attention task- Updating | 1 day
  Updating Attention
Miyake Executive Attention task-Shifting | 1 day
  Shifting Attention
Miyake Executive Attention task-Inhibition | 1 day
  Inhibition of attention
Working Memory Capacity | 1 day
  Estimate of working memory capacity based on behavioral performance

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Carlisle, PhD, Principal Investigator — Lehigh University
Locations (1):
- Lehigh University, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymous behavioral performance data will be available for other researchers upon request
Supporting Information: Study Protocol, Analytic Code
Time Frame: Upon publication of the work, for at least 5 years
Access Criteria: Request

REFERENCES:
- [Background] Arita JT, Carlisle NB, Woodman GF. Templates for rejection: configuring attention to ignore task-irrelevant features. J Exp Psychol Hum Percept Perform. 2012 Jun;38(3):580-4. doi: 10.1037/a0027885. Epub 2012 Apr 2. PMID 22468723
- [Background] Miyake A, Friedman NP, Emerson MJ, Witzki AH, Howerter A, Wager TD. The unity and diversity of executive functions and their contributions to complex "Frontal Lobe" tasks: a latent variable analysis. Cogn Psychol. 2000 Aug;41(1):49-100. doi: 10.1006/cogp.1999.0734. PMID 10945922